CLINICAL TRIAL: NCT03115801
Title: A Phase II Randomized Controlled Trial of Programmed Death -1/Programmed Death Ligand-1(PD-1/PDL-1) Axis Blockade Versus PD-1/PDL-1 Axis Blockade Plus Radiotherapy in Metastatic Genitourinary (Renal/Urothelial) Malignancies
Brief Title: A Phase II Randomized Trial of Immunotherapy Plus Radiotherapy in Metastatic Genitourinary Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1606017369
Record Dates: First submitted 2016-11-30; First posted 2017-04-14 (Actual); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Renal Cell Carcinoma; Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell | interventions — Nivolumab; Immunotherapy; atezolizumab; Radiation; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - immunotherapy alone (Active Comparator): Patients with Renal Cell carcinoma will receive Nivolumab alone Days 1, 15, 29, 43 and 57.
  Patients with Urothelial cancer will receive Atezolizumab or Pembrolizumab on Days 1, 22, 43 and 64.
  Interventions: Drug: Nivolumab; Drug: Atezolizumab; Drug: Pembrolizumab
- Arm B - Radiation & immunotherapy (Active Comparator): Radiation is given to one lesion, 30 Gy in 3 fractions of 10 Gy, every other day. On the day of radiation (Day 1) immunotherapy is administered and repeated on the scheduled days.
  Interventions: Drug: Nivolumab; Drug: Atezolizumab; Radiation: Radiation & immunotherapy

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be given to patients with renal cell carcinoma on days 1,15, 29, 43 and 57.
  Other Names: Immunotherapy
Drug: Atezolizumab — Atezolizumab will be given to patients with urothelial carcinoma on days 1,22,43,64.
  Other Names: Tecentriq
Radiation: Radiation & immunotherapy — Radiation is given to one lesion, 30 Gray (Gy) in 3 fractions of 10 Gy each. over a one week interval (with a minimum of 36hrs between each fraction). On the day of radiation (Day 1) immunotherapy is administered and repeated on the scheduled days. Patients will receive radiation on Day 1 and immunotherapy will be given ± 24hr from Day 1.
  Arms: Arm B - Radiation & immunotherapy
Drug: Pembrolizumab — Pembrolizumab will be given to patients with urothelial carcinoma on days 1,22,43,64.
  Other Names: Keytruda
  Arms: Arm A - immunotherapy alone

SUMMARY:
The trial is open to patients who have metastatic renal cell carcinoma/urothelial (bladder) carcinoma with at least 2 measurable sites of disease. All eligible patients will be randomly assigned to immunotherapy(nivolumab/atezolizumab/pembrolizumab) versus immunotherapy (nivolumab/atezolizumab/pembrolizumab) plus radiotherapy, 10 Gy x3 (conformally or by intensity modulation radiation therapy/Image-guided radiation therapy (IMRT/IGRT) to maximally spare normal tissue), to one of their measurable lesions.

DETAILED DESCRIPTION:
The trial is open to patients who have metastatic renal cell carcinoma/urothelial (bladder) carcinoma with at least 2 measurable sites of disease. All eligible patients will be randomly assigned to immunotherapy(nivolumab/atezolizumab/pembrolizumab) versus immunotherapy (nivolumab/atezolizumab/pembrolizumab) plus radiotherapy, 10 Gy x3 (conformally or by IMRT/IGRT to maximally spare normal tissue), to one of their measurable lesions. For patients assigned to the immunotherapy plus radiotherapy arm, immunotherapy treatment starts with the first radiotherapy fraction. Nivolumab will be given every 2 weeks for patients with metastatic renal cell cancer and atezolizumab/pembrolizumab will be given every 3 weeks for patients with metastatic urothelial cancer. Patients will be re-imaged at 9 week (year 1) or 12 week (years 2-3) intervals and evaluated for response (defined as an objective response of measurable metastatic sites outside the radiation field). This response will be evaluated with CT scans in non-irradiated measurable metastatic sites per RECIST version 1.1. Patients will continue to receive their respective immunotherapies for up to three years or until disease progression or until a dose limiting toxicity is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document;
2. Any prior therapy is permitted except prior therapy with PD1/PDL1 inhibitor.
3. Histologic diagnosis of metastatic renal cell carcinoma or urothelial cancer;
4. Patients must have at least 2 distinct measurable metastatic sites at least 1 cm or larger in their largest diameter per RECIST 1.1
5. Patients must have adequate organ and marrow function as defined by initial laboratory tests.
6. At least 2 weeks since last chemotherapy and 4 weeks since last immunotherapy treatment.
7. Performance status Eastern cooperative oncology group (ECOG) 0-1
8. Men and women, ages > 18 years of age.
9. Life expectancy > 3 months
10. Stable brain metastases for at least 4 weeks and not steroid dependent
11. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the study in such a manner that the risk of pregnancy is minimized. Should a woman become pregnant or suspect she is pregnant while she is enrolled in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. Patients having no lesions outside the field of radiation thus nullifying the ability to measure an abscopal effect;
2. Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix;
3. Autoimmune/auto inflammatory disease: Patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis];
4. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea;
5. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of PD-1/PDL-1 blocking antibody).
6. A history of prior treatment with PD-1/PDL-1blocking antibody;
7. Patients who have had immunotherapy within 4 weeks prior to entering the study.
8. Concomitant therapy with any of the following: interleukin -2 (IL-2), interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids;
9. Patients undergoing therapy with other investigational agents or other chemotherapy agents;
10. Women who:

    1. are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 8 weeks after cessation of study drug, or
    2. have a positive pregnancy test at baseline, or
    3. are pregnant or breastfeeding
11. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11; Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himanshu Nagar, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medicine - New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Immunotherapy Alone: Patients with Renal Cell carcinoma will receive Nivolumab alone Days 1, 15, 29, 43 and 57.
  Patients with Urothelial cancer will receive Atezolizumab or Pembrolizumab on Days 1, 22, 43 and 64.
  Nivolumab: Nivolumab will be given to patients with renal cell carcinoma on days 1,15, 29, 43 and 57.
  Atezolizumab: Atezolizumab will be given to patients with urothelial carcinoma on days 1,22,43,64.
  Pembrolizumab: Pembrolizumab will be given to patients with urothelial carcinoma on days 1,22,43,64.
Period: Overall Study
Arm/Group | Arm A - Immunotherapy Alone | Arm B - Radiation & Immunotherapy
Started | 4 | 2
Completed | 1 | 0
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Immunotherapy Alone | Arm B - Radiation & Immunotherapy | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Full Range); unit: years] | 56.25 [45 to 63] | 69 [55 to 83] | 60.5 [45 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Overall Response Rates of Immunotherapy Alone and of Immunotherapy Plus Radiotherapy (to a Single Metastatic Site).
Time Frame: from 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Immunotherapy Alone | Arm B - Radiation & Immunotherapy
Number analyzed (Participants) | 4 | 2
Participants | 4 | 2

2. Primary Outcome: Assess the Difference in Participants for the Best Overall Response Between the Two Groups, Immunotherapy Alone and of Immunotherapy Plus Radiotherapy(to a Single Metastatic Site).
Time Frame: from 96 weeks
Population: 3 participants on ARM A and 2 participants on ARM B could not be analyzed because they were withdrawn from the trial for disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Immunotherapy Alone | Arm B - Radiation & Immunotherapy
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

3. Secondary Outcome: Number of Participants With Progression Free Survival
Time Frame: from 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Immunotherapy Alone | Arm B - Radiation & Immunotherapy
Number analyzed (Participants) | 4 | 2
Participants | 1 | 0

4. Secondary Outcome: Number of Participants Who Experienced Toxicities Related to Immunotherapy and Immunotherapy Plus Radiotherapy Treatment Groups
Time Frame: from 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Immunotherapy Alone | Arm B - Radiation & Immunotherapy
Number analyzed (Participants) | 4 | 2
Participants | 1 | 1

5. Secondary Outcome: Participants Will be Measured for Overall Survival
Time Frame: from 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Immunotherapy Alone | Arm B - Radiation & Immunotherapy
Number analyzed (Participants) | 4 | 2
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm A - Immunotherapy Alone | Arm B - Radiation & Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/2
Other Adverse Events (participants affected / at risk) | 1/4 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Immunotherapy Alone (N=4) | Arm B - Radiation & Immunotherapy (N=2)
Abdominal Pain (Gastrointestinal disorders) | 1 (3) | 0 (0) — Left lower Quadrant Abdominal Pain with urination
Dyspnea on Exertion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) — Bilateral 2+ pitting edema (Grade 2) and shortness of breath (Grade 2) were observed.
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) — Right hip fracture
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Hyperglycemia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Immunotherapy Alone (N=4) | Arm B - Radiation & Immunotherapy (N=2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Elevated Alkaline Phosphate (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Intermittent discomfort in the right buttock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03115801/Prot_SAP_000.pdf